CLINICAL TRIAL: NCT01927991
Title: Internet-based Self-help for Tinnitus: The Role of Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Cornelia Weise, Dr. rer. nat., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Titus2
Record Dates: First submitted 2013-08-17; First posted 2013-08-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Tinnitus
Keywords: tinnitus; cognitive behavioural therapy; internet treatment
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iCBT with therapeutic support (Experimental): Participants work with the online self-help and receive additional therapeutic support on demand
  Interventions: Behavioral: iCBT (internet-based, cognitive-behavioural therapy)
- iCBT without therapeutic support (Active Comparator): Participants work with the online self-help on their own and do not receive additional therapeutic support
  Interventions: Behavioral: iCBT (internet-based, cognitive-behavioural therapy)

INTERVENTIONS:
Behavioral: iCBT (internet-based, cognitive-behavioural therapy) — The intervention is based on cognitive-behavioural therapy (CBT) and is offered as a self-help and provided over the internet. Participants work on their own on different modules which give information about tinnitus and the associated symptoms and provide instructions for practical exercises.

SUMMARY:
Internet-based cognitive behavioural self-help (iCBT) has become increasingly popular to provide psychotherapy. For several psychological and psychosomatic disorders, treatment efficacy was shown. Previously, iCBT has also been applied to patients suffering from tinnitus and results show significant and long-term stable improvements in tinnitus distress. However, the role of therapeutic support in iCBT has not been thoroughly investigated. Previous results suggest that iCBT without therapeutic support is less effective and leads to higher dropout rates than therapist-guided iCBT. The aim of the randomized controlled trial is thus to investigate the role of therapeutic support in an iCBT for tinnitus sufferers.

ELIGIBILITY:
Inclusion Criteria:

* tinnitus duration of more than 6 months
* severe or most severe tinnitus distress
* age of at least 18 years
* fluent in German

Exclusion Criteria:

* psychosis, severe psychological disorder, risk for suicide
* prior participation in associated study
* medical disorder as reason for tinnitus, i.e. morbus ménière

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in tinnitus distress | 1 year; pre, post, 6-mo-follow-up
  Assessment of tinnitus distress with the Tinnitus Handicap Inventory (THI) and the Mini-Tinnitus Questionnaire (Mini-TQ)
  Newman, C. W., Jacobson, G. P., & Spitzer, J. B. (1996). Development of the Tinnitus Handicap Inventory. Arch Otolaryngol Head Neck Surg, 122(2), 143-148.
  Hiller, W., & Goebel, G. (2004). Rapid assessment of tinnitus-related psychological distress using the Mini-TQ. Int J Audiol, 43(10), 600-604.

SECONDARY OUTCOMES:
Change in depressive Symptoms | 1 year; pre, post, 6mo-follow-up
  Assessment of depressive symptoms with the Patient Health Questionnaire (PHQ-9) and the Hospital Anxiety and Depression Scale (HADS)
  Kroenke, K., Spitzer, R. L., & Williams, J. B. W. (2001). The PHQ-9: Validity of a brief depression severity measure. J Gen Intern Med, 16(9), 606-613. 10.1046/j.1525-1497.2001.016009606.x
  Zigmond, A. S., & Snaith, R. P. (1983). The hospital anxiety and depression scale. Acta Psychiatr Scand, 67(6), 361-370.
Change in tinnitus-related thoughts | 1 year; pre, post, 6mo-follow-up
  Assessment of dysfunctional tinnitus-related thoughts with the Tinnitus Cognitions Scale (T-Cog)
  Hiller, W., & Haerkötter, C. (2005). Does sound stimulation have additive effects on cognitive-behavioral treatment of chronic tinnitus? Behav Res Ther, 43(5), 595-612.
Change of tinnitus acceptance | 1 year; pre, post, 6mo-follow-up
  Assessment of tinnitus acceptance with the Tinnitus Acceptance Questionnaire (TAQ)
  Weise, C., Kleinstauber, M., Hesser, H., Westin, V. Z., & Andersson, G. (2013). Acceptance of tinnitus: validation of the tinnitus acceptance questionnaire. Cognitive Behaviour Therapy, 42(2), 100-115. 10.1080/16506073.2013.781670

OTHER OUTCOMES:
Screening of psychiatric symptoms | Pre-Treatment
  Assessment of psychiatric disorders at pre-treatment
  Donker, T., van Straten, A., Marks, I., & Cuijpers, P. (2009). A Brief Web-Based Screening Questionnaire for Common Mental Disorders: Development and Validation. Journal of Medical Internet Research, 11(3), Artn E19. Doi 10.2196/Jmir.1134

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Weise, Dr., Principal Investigator — Philipps-University Marburg, Dept. of Psychology, Division of Clinical Psychology and Psychotherapy
Locations (1):
- Philipps University Marburg, Dept. of Psychology, Division of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany